CLINICAL TRIAL: NCT06696196
Title: Validation of Sleep Monitoring Algorithm Based on Smart Watches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201503059RSA
Record Dates: First submitted 2023-06-29; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Polysomnography; sleep staging; sleep efficiency; wearable devices; smart watches
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- smart watch (Experimental): This study will use a prototype (MediaTek Sleep Watch) to acquire PPG, body movements, skin temperature, and skin conductance to validate the algorithm of sleep staging and sleep efficiency assessment. PSG will be used as gold standard for statistical analysis.
  Interventions: Device: smart watches(wearable devices)

INTERVENTIONS:
Device: smart watches(wearable devices) — Participants will be asked to wear two smart watches simultaneously. The first smart watch is a dedicated prototype for validating algorithm developed by MediaTek. The second smart watch is Basis Peak. These watches are going to acquire PPG, body movements, skin temperature, and skin conductance.

SUMMARY:
In recent years, wearable devices are booming to enable not only the health monitoring but also the sleep efficiency assessment. To validate the algorithm of sleep staging and efficiency, this study will use a dedicated prototype to acquire photoplethysmogram (PPG), body movements, skin temperature, and galvanic skin response by recruiting 35 subjects. PSG will be used as gold standard for statistical analysi.

DETAILED DESCRIPTION:
Sleep efficiency has a great impact on the performance of work and learning during the day. If persons lack of sleep for a long time, they might be prone to memory loss and emotional instability. Traditionally, polysomnography (PSG) has been proved as golden results to assess the sleep efficiency. However, to accomplish the assessment, subjects are asked to sleep in a certified sleep laboratory or a sleep centers for nights. Under the supervision of nurses, subjects are put many adhesive electrodes on the body and connect wires to PSG, which causes discomfort. In recent years, wearable devices are booming to enable not only the health monitoring but also the sleep efficiency assessment. To validate the algorithm of sleep staging and efficiency, this study will use a dedicated prototype to acquire photoplethysmogram (PPG), body movements, skin temperature, and galvanic skin response by recruiting 35 subjects. PSG will be used as gold standard for statistical analysi.

ELIGIBILITY:
Inclusion Criteria:

1. Forty male or female subjects are recruited from those visiting Department of Medicine for health check up
2. Subjects aged 20 to 65

Exclusion Criteria:

1. Refuse to participate
2. Arrhythmia
3. Active infection
4. Active neurologic event
5. Shift worker
6. Substance abuse
7. Fitted with implantable medical electronics, such as cardiac pacemakers and defibrillators

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
sleep stages derived from smartwatch | 12 months
  Comparing sleep stages detected by a smartwatch(hh:mm) with the sleep stages of an overnight PSG(N1 (%), N2 (%), N3 (%), REM(%), Arousal index (/h) to validate the effectiveness of the smartwatch.

SECONDARY OUTCOMES:
sleep efficiency derived from smartwatch | 12 months
  Comparing sleep efficiency(%) detected by a smartwatch with the sleep efficiency(%) from an overnight PSG to validate the effectiveness of the smartwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Lin Lee, M.D., PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No